CLINICAL TRIAL: NCT03206541
Title: Neurovirus Emerging in the Americas Study (NEAS): Neurologic Manifestations of the Arbovirus Dengue, Chikungunya and Zika Infections in Colombia
Brief Title: Neurologic Manifestations of the Arbovirus Infection in Colombia
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Universidad del Valle, Colombia (Other); ZikaPLAN (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00093149
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Encephalitis; Myelitis; Guillain-Barre Syndrome; Cranial Nerve Palsies; Meningitis; Zika Virus Infection; Dengue (Virus); Fever, Sandfly; Chikungunya Fever
Keywords: Neurological syndromes; Arbovirus infection
MeSH Terms: conditions — Encephalitis; Myelitis; Guillain-Barre Syndrome; Cranial Nerve Diseases; Meningitis; Zika Virus Infection; Dengue; Virus Diseases; Fever; Chikungunya Fever; Arbovirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — The study will retain blood (serum and plasma), urine, spinal fluid and saliva for cases and controls according to the protocol. The samples will remain in the core laboratory at UV and some of them will be shared with the JHU team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: The cases are defined as individuals that present with new onset of a neurological syndrome of unknown etiology, including but not limited to encephalitis, myelitis, meningitis, polyneuropathy/Guillain-Barre syndrome and cranial nerve involvement.
- Controls: There are two age-matched control groups:
  1. Household controls that have lived with the case for at least three months before the onset of neurological symptoms.
  2. Controls with a febrile syndrome of unknown etiology that do not present neurological involvement and is recruited in the same center as the case.

SUMMARY:
This is a multi-center case-control study that aims to define the association between the exposure to an arbovirus infection and the development of a neurological syndrome in patients from Colombia. The study makes part of the Neurovirus Emerging in the Americas Study (NEAS) that is a collaborative effort that looks to combine the efforts of researchers, healthcare providers and patients in Colombia to establish a comprehensive registry of the clinical, radiological and laboratory profile of patients with new onset of neurological diseases associated mosquito-borne viruses, known as arboviruses.

DETAILED DESCRIPTION:
NEAS is led by Dr. Carlos Pardo-Villamizar at Johns Hopkins University (JHU) and Drs. Beatriz Parra and Lyda Osorio at Universidad del Valle (UV) in Colombia. They have established a collaborative network with physicians, neurologists and experts in microbiology and epidemiology in that country. NEAS is actively recruiting patients in seven university-based hospitals in five Colombian cities. The protocol of the study has been approved in each of the participating centers.

NEAS prospective case-control study aims to define the association between the exposure to arbovirus (Zika, Dengue and Chikungunya) and the development of a neurological syndrome in patients from Colombia, a country with endemic transmission of arbovirus. The cases are defined as individuals that present with new onset of a neurological syndrome of unknown etiology, including but not limited to encephalitis, myelitis, meningitis, polyneuropathy/Guillain-Barre syndrome and cranial nerve involvement. There are two age-matched control groups: 1) household controls and 2) controls with a febrile syndrome of unknown etiology that do not present neurological involvement. The estimated sample size in the study is 50 participants in each group (cases and controls 1 and 2). The time to collect the complete sample size is between 12-24 months, and depends on the local incidence of cases.

Each center has a coordinator team that includes a neurologist, a physician - neurology or internal medicine resident -, and a research coordinator. The team is constantly screening the patients admitted to the center. The patients that fulfill the criteria for cases or controls are approached by the research coordinator who is in charge to inform the participant about the study and complete the informed consent. Then, the medical team perform the neurological evaluation, including the history and the physical exam according to the NEAS forms. Samples of blood and urine are collected in all participants. If a lumbar puncture is done as part of the standard of care, spinal fluid is also collected. Based on resources availability, the participants are followed every week for a 4-week period and in each visit a clinical assessment and sample collection are completed.

Demographic and clinical information, laboratory and imaging results are stored in a secured web-based database in the platform REDcap,based at JHU. Each center has a unique combination of a username and a password to enter the database and include the information of each participant in real time. Each center has access to the included information by the same center and no by other centers. Standardized forms (NEAS forms) were created by the study team that include relevant information necessary to achieved the aims of this study and guarantee the data consistency. Laboratory testing and imaging results are obtained from the medical records. A permanent monitoring of the data base is done by the teams at JHU and UV.

After the samples are collected they are shipped to the study core laboratory located at UV (Dr. Beatriz Parra). Each center has been trained in the correct handling, processing, and shipping of the samples. Once the samples are in the core laboratory, they are aliquoted and stored. Blood, urine and spinal fluid are tested by Real Time/Reverse Transcriptase (RT)- Polymerase Chain Reaction (PCR) for the presence of viral RNA (Ribonucleic Acid) of Zika virus and Dengue virus. Serum and spinal fluid are tested by ELISA for the detection of anti-flavivirus IgM and IgG. The results are shared with the local study team and with the medical team taking care of the participant. In addition, aliquots of samples are sent to JHU for additional immunological and virological assessments (Dr. Carlos Pardo-Vllamizar).

Standard Operative Procedures (SOP) have been created for patient recruitment and consent, REDcap data entering, and biosamples process and shipment. The statistical analysis will be done by epidemiologists at UV (Dr. Lyda Osorio) and it will include frequency measures and central tendency measures of the variables. The measure of the strength of association will be done using Odds ratio and confidence intervals.

DATA DICTIONARY

The variables are divided in three categories: demographic, clinical and laboratory. The most relevant variables collected in the study are described below.

Demographic variables:

* Case: Case definition
* Type of control: Control definition
* Fulfillment of the inclusion criteria: Fulfillment of the inclusion criteria established by the protocol
* Gender: Sexual phenotype of the participant supported by the medical records or ID
* Age: Participant's age according to the medical records or ID
* Race: Phenotype reported by the participant
* City of residence: Place where has mainly been in the last 3 months
* City of report: Place where the participant is recruited to the study

Clinical variables:

* General symptoms: Clinical manifestations consistent with decrease in the normal health shape of the participant
* Onset of general symptoms: Date of the onset of general symptoms
* Neurological symptoms: Clinical manifestations reflecting an abnormal functioning of the nervous system
* Temporal profile: Time (in days) between the onset of general symptoms and neurological symptoms
* Visit to endemic regions: History of have visited during the last 4 weeks regions with current local transmission of Zika, Dengue and/or Chikungunya virus
* Past medical history: History of a disease diagnosed by the doctor or reported in the medical records during the past year
* Family history: Diseases suffered by first or second consanguinity degree relatives diagnosed by the doctor or reported in the medical records
* Recent vaccination: History of vaccination during the past 4 weeks before the onset of the neurological symptoms
* Recent infectious disease: History of an infectious disease during the past 4 weeks before the onset of the neurological symptoms
* Recent surgical procedure: History of a major surgical procedure during the past 4 weeks before the onset of the neurological symptoms
* Date of physical exam: Date when physical exam was completed by the study team
* Mental status: Range of own/outer consciousness
* Orientation: Awareness of time, place and person
* Dysarthria: Word articulation dysfunction secondary to a motor pathways damage
* Attention deficit: Inability to selectively concentrate in an specific portion of the information
* Cranial nerves abnormalities: Compromise of one/more of the cranial nerves detected on the physical exam
* Muscle strength: Amount of strength done by a muscle against resistance
* Deep tendon reflexes: Extension secondary to a deep tendon stimulus
* Sensory deficit: Absence or abnormality in the sensory function
* Romberg sign: Clinical sign suggesting sensory ataxia, secondary to dorsal columns abnormalities
* Ataxia: Abnormal muscle coordination during voluntary movements
* Muscle tone: Muscle resistance against passive movement
* Urinary retention: Inability to complete bladder emptiness
* Low rectal muscle tone: Decrease in the strength of the rectal sphincter
* Abnormal movements: No voluntary movements, without purpose, secondary to a neurological dysfunction
* Respiratory failure: Inability to perform an efficient gas exchange or to maintain normal levels of oxygen and/or carbon dioxide
* Autonomic dysfunction: Abnormalities in the autonomic nervous system
* Electromyography: Electrophysiological study of the muscle activity
* Electroencephalogram: Electrophysiological study of the brain conduction
* Brain MRI: Imaging study of the brain
* Spinal cord MRI: Imaging study of the spinal cord
* Rankin score: Functional scale for patients with neurological disorders
* ASIA scale: Severity of spinal cord lesion

Laboratory variables:

* Blood analysis: Include white blood cells count, platelets, hemoglobin, hematocrit and liver function enzymes.
* Spinal fluid analysis: Includes leukocytes, glucose, proteins, red blood cells, oligoclonal bands, cultures, herpes virus PCR.
* Virological analysis: Includes detection or absence of detection of IgM and IgG by ELISA, and the RNA by RT-PCR for Zika virus, Dengue virus and Chikungunya virus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Case or control definition
* Informed consent or assent

Exclusion Criteria:

* Known etiology for the acute neurological disorders
* History of known neurological syndrome

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes males and females over 8 years of age at risk of being infected by Dengue, Chikungunya or Zika viruses.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Neurological outcomes in arbovirus infections | 12-24 months
  Number of patients with neurological syndromes that have evidence of acute infection by Zika, Dengue or Chikungunya viruses assessed by IgM serology or polymerase chain reaction

SECONDARY OUTCOMES:
Viral genotype | 24-36 months
  Number of strains of Zika, Dengue and Chikungunya viruses assessed by genome sequencing
Immune response | 24-36 months
  Cellular immune response assessed by T-lymphocyte profiling in patients with confirmed arbovirus infection with and without neurological syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Pardo-Villamizar, MD, Principal Investigator — Johns Hopkins University; Beatriz Parra, PhD, Principal Investigator — Universidad del Valle; Lyda Osorio, PhD, Principal Investigator — Universidad del Valle
Locations (8):
- Colombia (8):
  - Clinica Leon XIII, Medellín, Antioquia
  - Neuroclinica, Medellín, Antioquia
  - Clinica La Misericordia Internacional, Barranquilla, Atlántico
  - Hospital Universitario de Narino, Pasto, Departamento de Nariño
  - Clinica Medilaser, Neiva, Huila Department
  - Hospital Universitario de Neiva, Neiva, Huila Department
  - Hospital Universitario Erasmo Meoz, Cúcuta, Norte de Santander Department
  - Hospital Universitario del Valle, Cali, Valle del Cauca Department

IPD SHARING:
Plan to Share IPD: Yes
NEAS is part of the ZikaPLAN, which is a consortium led by the European Community. There is a plan of sharing information with other collaborators within the consortium. The information will include demographic information, laboratory results and neurological physical exam. No identifiers will be shared. The information will be obtained through the ongoing recruitment of patients. We plan to share the first set of information during the second semester of 2017.

REFERENCES:
- [Background] Munoz LS, Barreras P, Pardo CA. Zika Virus-Associated Neurological Disease in the Adult: Guillain-Barre Syndrome, Encephalitis, and Myelitis. Semin Reprod Med. 2016 Sep;34(5):273-279. doi: 10.1055/s-0036-1592066. Epub 2016 Sep 9. PMID 27612158
- [Background] Rowland A, Washington CI, Sheffield JS, Pardo-Villamizar CA, Segars JH. Zika virus infection in semen: a call to action and research. J Assist Reprod Genet. 2016 Apr;33(4):435-7. doi: 10.1007/s10815-016-0684-6. Epub 2016 Mar 5. No abstract available. PMID 26945753
- [Result] Parra B, Lizarazo J, Jimenez-Arango JA, Zea-Vera AF, Gonzalez-Manrique G, Vargas J, Angarita JA, Zuniga G, Lopez-Gonzalez R, Beltran CL, Rizcala KH, Morales MT, Pacheco O, Ospina ML, Kumar A, Cornblath DR, Munoz LS, Osorio L, Barreras P, Pardo CA. Guillain-Barre Syndrome Associated with Zika Virus Infection in Colombia. N Engl J Med. 2016 Oct 20;375(16):1513-1523. doi: 10.1056/NEJMoa1605564. Epub 2016 Oct 5. PMID 27705091
- [Result] Zea-Vera AF, Parra B. Zika virus (ZIKV) infection related with immune thrombocytopenic purpura (ITP) exacerbation and antinuclear antibody positivity. Lupus. 2017 Jul;26(8):890-892. doi: 10.1177/0961203316671816. Epub 2016 Sep 30. PMID 27694629